CLINICAL TRIAL: NCT05561192
Title: Effects of Insertion of Diaphragmatic Breathing Exercises, Cardiorespiratory and Strength Exercises, and Cooperative Sports Activities During Physical Education Classes on Anxiety and Depression Symptoms in Adolescents
Brief Title: Effects of Inserting Exercises During Physical Education Classes on Anxiety and Depression Symptoms in Adolescents
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Federal University of Pelotas (Other)
Responsible Party: Principal Investigator, Gabriel Gustavo Bergmann, Director, Federal University of Pelotas
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Int_IFSUL
Record Dates: First submitted 2022-08-23; First posted 2022-09-30 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Depressive Symptoms; Anxiety Symptoms
Keywords: depressive symptoms; anxiety symptoms; physical education; school; intervention; breathing exercises; physical exercises; cooperative sports activities
MeSH Terms: conditions — Depression; Anxiety Disorders; Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Given the nature of this project, it will not be possible to blind the samples (classes) participating in the study due to the clarity of the intervention process (diaphragmatic breathing exercises, cardiorespiratory and strength exercises and cooperative sports activities) not even from teachers or external applicators. However, it is important to note that there will be blinding of the process within the following points:
  * Applicators of the instruments (questionnaires) and evaluators teachers, who will carry out the anthropometric evaluations of the subjects;
  * Tabulation and data analysis;
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- diaphragmatic breathing exercises group (Experimental): Intervention with diaphragmatic breathing exercises will take place in the last 15 minutes of Physical Education classes, focusing on diaphragmatic breathing. This breathing is also characterized by reducing the respiratory cycle or rate, and it can use the count of seconds in a progressive way, either in the inhalation through the nose while the abdomen expands, in the support or blockage or also called pause, and finally in the expiration, also performed by the nostrils. The creation of an inhalation and exhalation pattern becomes important as it has a direct relationship with the reduction of the activities of the sympathetic nervous system and the increase of the activity of the parasympathetic nervous system, also influencing the motor activities, the brain mass, the quality of the sleep and the attenuation of stressors.
  Interventions: Other: Diaphragmatic breathing exercises
- Cardiorespiratory and strength exercise group (Experimental): Intervention with cardiorespiratory and strength physical exercises will always occur in the first 15 minutes of each class. Cardiorespiratory exercises and localized muscular resistance will be developed involving all muscle groups, adapted to the materials and school equipment available. The exercises developed will be primarily calisthenics, to facilitate a possible replication within the school environment. A circuit with 4 stations will be elaborated, where one station will offer a cardiorespiratory stimulus, containing the following exercises: jumping jacks, jumping rope, stationary running, going up and down steps and burpees. The other three stations will be composed of localized muscular resistance exercises, involving lower limbs (squat, lunge and isometric chair), upper limbs (flexion) and trunk (abdominal).
  The time of execution of the exercises in each station will be of 1 minute.
  Interventions: Other: Cardiorespiratory and strength exercise
- Cooperative sports activities group (Experimental): The intervention of cooperative sports activities that will integrate the physical education class will be based on the cooperative learning model and elaborated through the aforementioned points. Intervention sessions will last 20 minutes, being held during the main part of the class. Activities will be planned that prioritize reflection, thinking and sharing of ideas among students, by proposing challenges within the sport. For example, how to get out of a certain type of marking within a game, or in the case of cooperative games, with the principle that students cooperate with each other to solve a proposed challenge (for example, how long a team can remain dominating the volleyball without it falling to the ground?).
  Interventions: Other: Cooperative sports activities group
- Comparator Group (Active Comparator): The classes that will form the comparator group will carry out the Physical Education classes according to the planning previously prepared by the professors of the discipline and that are already part of the syllabus of the semester and/or the school year of the classes. These contents, within the proposal of the two schools, are already consolidated and are centered on the teaching of sport through methodologies aimed at a pedagogical proposal mostly analytical, partial or characterized by the traditional model (technicist model). In these classes, the activities are practiced through the model of direct instruction of teaching, where the teacher acts as the main figure of the teaching-learning process.
  Interventions: Other: Traditional physical education class

INTERVENTIONS:
Other: Diaphragmatic breathing exercises — The initial proposal is for the first week to be adaptive, that is, learning to perform the exercises freely. During this period, students will be able to experience the activities and solve any doubts, as well as understand the process of a respiratory cycle, in which they will be initiated through a cycle of 12 times per minute. In the second and third weeks, the exercises will consist of 10 breathing cycles per minute (complete cycle consisting of 6 seconds, 2:2:2). It is important to note that each cycle contains the inspiration time, brief pause and expiration time in seconds. In the last week, each cycle will last 16 seconds, consisting of 4 seconds of inspiration, 4 seconds of pause and 8 seconds of expiration (4:4:8). Thus, the objective is to reduce the number of respiratory cycles per minute, as the intervention progresses.
  Arms: diaphragmatic breathing exercises group
Other: Cardiorespiratory and strength exercise — During the first two weeks, students will complete two laps of the circuit, with a 15-second break between one station and another and a 1-minute break between one lap and another. These first two weeks will focus on adaptation and technical learning of the exercises to be performed. From the third to the sixth week, one lap will be added to the circuit, totaling three laps, maintaining the aforementioned intervals. From week 7 to week 12, progressions will be carried out, reducing the interval time between one lap and another on the circuit to 30 seconds. For the purpose of controlling the intensity of the exercise, a subjective perception of effort scale will be used, composed of values from 1 to 10, the first being equivalent to "very light" effort activity, and ten, equivalent to "maximum effort activity".
  Arms: Cardiorespiratory and strength exercise group
Other: Cooperative sports activities group — Intervention with cooperative sports activities will be based on the pedagogical model for teaching sports called "Cooperative Learning" or "Cooperative Learning". This pedagogical model has some predominant characteristics, such as student learning occurring with and through other students, through an approach that facilitates and enhances positive interdependence, where teachers and students act as co-learners. Thus, this teaching model encompasses two key points of cooperative learning: promoting interaction between students and interaction between students and teachers.
  Also, in the planning of intervention classes with sports, the five points described as fundamental for learning to be considered cooperative will be considered. These are: face-to-face interaction, positive interdependence, individual responsibility, group processing, and social skills.
  Arms: Cooperative sports activities group
Other: Traditional physical education class — The comparator group will take physical education classes normally, following the traditional menu in the discipline, without changes in the conduct of activities.
  Arms: Comparator Group

SUMMARY:
The main objective of this project will be to verify if the insertion of diaphragmatic, cardiorespiratory and strength breathing exercises and cooperative sports activities in Physical Education classes, during a period of 12 weeks, may be able to modify the scores of symptoms of anxiety and depression in adolescent students. As secondary objectives, this project will seek to verify which of the interventions will provide the greatest reductions in students' anxiety and depression symptoms, as well as analyze their effects on other health indicators, also verifying if a greater volume of sessions can provide additional benefits to mental health. when compared to a smaller volume. This is an experimental study, of the randomized clinical trial (RCT) type. The target population will be adolescent students (14 to 19 years old) from the Federal Institute Sul-rio-grandense (IFSul) on the Bagé and Pelotas campuses. A total of 16 classes will compose the sample. The classes that have the Physical Education (PE) curriculum component in their schedule will be listed and randomized in relation to the comparator group (CG) and to the three different intervention protocols: diaphragmatic breathing exercises (intervention group 1 or GI-1), physical exercises cardiorespiratory and strength activities (intervention group 2 or GI-2) and cooperative sports activities (intervention group 3 or GI-3). The application of these interventions will occur during PE classes, twice a week at Campus Bagé and three times a week at Campus Pelotas. Interventions will last 15 minutes in groups GI-1 and GI-2, and 20 minutes in GI-3. Before the start of the intervention, baseline assessments will be carried out, consisting of primary outcomes (symptoms of anxiety and depression) and secondary outcomes (self-concept, quality of life, sleep indicators, self-perception of physical fitness, cognitive failures, strength and cardiorespiratory fitness). The groups will be compared regarding the characteristics collected at baseline and after the 12th week of intervention. The Generalized Estimating Equations (GEE) and the post-hoc Bonferroni test will be used to compare the moments (pre and post-intervention) between the groups and to identify the group*moment interaction. Analyzes will be performed by protocol and by intention to treat. The significance coefficient adopted will be p<0.05.

DETAILED DESCRIPTION:
General objective To evaluate the effects of interventions with diaphragmatic breathing exercises, cardiorespiratory and strength exercises, and cooperative sports practices on anxiety and depression symptoms in adolescents during high school physical education classes.

Specific

* To compare the effects of interventions with diaphragmatic breathing exercises, cardiorespiratory and strength exercises and cooperative sports practices on students' anxiety and depression symptoms;
* Analyze the effect and compare the interventions carried out in relation to the different health indicators: Quality of life, Sleep indicators, Self-concept, Self-perception of physical fitness, Cognitive failures, Strength (maximum, resistance and power) and Cardiorespiratory fitness;
* Verify and compare the effect of interventions with different weekly volumes (twice a week and three times a week) on students' anxiety and depression symptoms, as well as on the secondary outcomes analyzed.

Target Population and Sample The target population will be integrated high school students from the Federal Institutes of Rio Grande do Sul. The study sample will be composed of students (14 to 19 years old) of the integrated high school of the Federal Institutes of Sul-rio-grandense (IFSul) Campus Pelotas and Bagé.

Sample characterization variables demographic indicators

* Gender identity;
* Age;
* Marital status;
* Skin color.

Socioeconomic indicators

* Socioeconomic level through monthly family income (BRL);
* Campus you study;
* Course and year/semester attended.

Anthropometric indicators

* Body mass (kilograms);
* Height (meters);
* Body Mass Index (BMI).

Clinical indicators

* Previous clinical diagnosis of anxiety or depression disorder in the student;
* History of any diagnosed anxiety disorder in the family (father/mother);
* History of any diagnosed depressive disorder in the family (father/mother);
* Use of continuous use of anxiolytic;
* Use of continuous use antidepressant;
* Need for psychological or psychiatric follow-up in the last 12 months;
* Current psychological or psychiatric follow-up.

Control variables

* Level of physical activity;
* Screen time;
* Habitual practice of physical activity.

Instruments Anxiety Symptoms: Anxiety symptoms will be collected using the General Anxiety Disorder-7 (GAD-7) instrument. The General Anxiety Disorder-7 (GAD-7) instrument seeks to assess and monitor anxiety symptoms.

Depressive symptoms: To assess depressive symptoms, the Patient Health Questionnaire-9 (PHQ-9) instrument will be used, which seeks to assess and monitor depressive symptoms.

Self-concept: This assessment will be obtained through the Multidimensional Self-Concept Scale (AF-5).

Quality of Life: For the assessment of quality of life, the instrument World Health Organization Quality of Life (WHOQOL) abbreviated version, proposed by the World Health Organization.

Self-perception of physical fitness: For the assessment the self-perception of physical fitness will be used the Physical Fitness Questionnaire (International Fitness Scale - IFIS).

Cognitive Failures: For the assessment the cognitive failures will be used the Cognitive Failures Questionnaire (CFQ).

Physical activity level: The instrument to measure physical activity will be the International Physical Activity Questionnaire (IPAQ), short version, proposed by the World Health Organization (WHO) and the Center for Disease Control and Prevention (CDC).

Screen time: The variable "sedentary screen time" during leisure will be evaluated by the time of hours per day in which the person uses television, computer, tablet, cell phone and video game, in the face of a posture that implies low energy expenditure , such as sitting or lying down.

Habitual practice of physical activity: This variable will be analyzed through simple questions, such as "Do you currently practice any type of physical activity regularly? If yes, describe which one(s)."; "Is this physical activity performed under the supervision of a professional (teacher/technician)?"; "Where do you practice this physical activity?"; "Do you participate in competitions with this physical activity?". The mentioned questions aim to investigate the habitual practice of physical activities, the type, presence of supervision, location and purpose of these practices.

Body Mass Index: The body mass index (BMI) will be calculated by the body mass (Kg) measured, divided by the height (in meters) squared.

Strength: The maximum muscular strength will be measured through the handgrip strength by a hydraulic dynamometer.

The power of lower limbs will be evaluated through the horizontal jump test.

Endurance strength will be measured by the 1-minute abdominal endurance test.

Cardiorespiratory fitness: Cardiorespiratory fitness will be assessed through the 20m back and forth test.

Demographic variables

To collect information regarding demographic variables, the respondent will be asked to do the following:

* Tick one of the options in the gender question.
* Fill in your current age in complete years;
* Tick one of the options in the marital status question;
* Tick one of the options in the skin color question.

Socioeconomic indicators

For the collection of information regarding the socioeconomic variables, the respondent will be asked the following:

* Fill in the total monthly family income (BRL);
* Fill in the campus where you study (Bagé or Pelotas);
* Fill in the year or semester of the course you are enrolled and attending. The courses are as follows: agriculture, information technology, visual communication, interior design, buildings, electromechanics, electronics, electrotechnical and chemistry.

Anthropometric indicators To verify the anthropometric indicators, measurements of body weight (in kg) and height (in cm) will be performed. Body weight will be obtained using a scale, and students will be instructed to wear light clothes and be barefoot. Height will be measured using a stadiometer attached to the aforementioned scale.

Clinical indicators Student or family history of anxiety or depression disorder (parent); The history of anxiety or depression disorder in the student or in the father and/or mother will be collected through a closed question in which it will be asked if the student has a clinical diagnosis of anxiety or depression disorder and if any family member (father/mother) is or has been diagnosed with some form of anxiety disorder or depressive disorder. If positive in any of the questions, specify which disorder.

Drug intake Continuous use drugs will be collected through a closed question in which the person will be asked if the person uses anxiolytic or antidepressant drugs of continuous use and, if so, the name of these drugs and the doses ingested.

Psychological or psychiatric support Two questions will be made available about the need for some psychological or psychiatric follow-up. The first addressing whether there was psychological or psychiatric follow-up in the last 12 months and the second whether this service is currently needed.

Data analysis Initially, the numerical variables will be analyzed in relation to the normality of their distributions using the Shapiro-Wilk test. The description of numerical variables will be performed by the mean and standard deviation (sd) or median and interquartile intervals. The description of the categorical variables will be performed by the absolute (n) and relative (%) frequencies. To compare the characterization variables between the groups, ANOVA and the chi-square test will be used for numerical and categorical variables, respectively. Generalized Estimating Equations (GEE) and Bonferroni's post-hoc test will be used to compare moments (pre and post-intervention) and between groups to identify the group*moment interaction. Analyzes will be performed by intention to treat and by protocol. In intention-to-treat analyses, all participants will be included. Participants who do not present consistent data in at least one of the moments (pre and/or post-intervention) and those students who present any of the aforementioned exclusion criteria will be removed from the protocol analyses. It will also be verified the effect size amplitude through Cohen's "d", obtaining the classification: insignificant (≤0.19) small (0.20 to 0.49); medium (0.50 to 0.79); large (0.80 to 1.29) and very large (≥1.30), according to Cohen (1988) and Rosenthal (1996). The significance level adopted will be 5% for all statistical analyses.

ELIGIBILITY:
Inclusion Criteria:

* Students who are regularly enrolled and attending Physical Education classes at the integrated high school of IFSul Campus Bagé and Pelotas;

Exclusion Criterias:

* Students under 14 years of age or over 19 years;
* Students with any physical or health limitation that prevents the execution of practical activities, as well as those supported by a medical certificate;
* Students who do not reach the minimum attendance of 75% in physical education classes;
* Students who present a clinical diagnosis of anxiety or depression;
* Students who use medication for anxiety or depression;
* Students who are currently undergoing psychiatric or psychological follow-up or who have performed this professional follow-up in the last 12 months.

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 320 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Depressive Symptoms | Depressive symptoms will be assessed at week 0 (pre-intervention) and week 13 (post-intervention).
  Depressive symptoms will be assessed using the PHQ-9 instrument. The instrument measurements range from 0 to 27 points, with values greater than 10 indicating depressive symptoms.
Change in Anxiety Symptoms | Anxiety symptoms will be assessed at week 0 (pre-intervention) and week 13 (post-intervention).
  Anxiety symptoms will be assessed using the GAD-7 instrument. The instrument measurements range from 0 to 21 points, with values greater than 10 indicating anxiety symptoms.

SECONDARY OUTCOMES:
Change in Self-concept | Self-concept will be assessed at week 0 (pre-intervention) and week 13 (post-intervention).
  This assessment will be obtained through the Multidimensional Self-Concept Scale (AF-5). The instrument consists of 24 items and the result will be verified through the sum of each of the answered items, and the higher the total score, the greater the assessment of self-concept.
Change in Quality of Life | Quality of life will be assessed at week 0 (pre-intervention) and week 13 (post-intervention).
  This assessment will be obtained through the WHOQoL (World Health Organization-Quality of Life- Brief). The instrument consists of 26 items. The results will be transformed into a linear scale, which may vary from 0 to 100, and the higher the result found, the greater the perception of quality of life of the subject.
Change in Sleep Indicators | Sleep indicators will be assessed at week 0 (pre-intervention) and week 13 (post-intervention).
  This assessment will be obtained through the Pittsburgh Sleep Quality Index (PSQI). The instrument consists of 19 self-administered questions. The results are obtained by a global score that varies from 0 to 21 points and the higher the score, the worse the sleep quality.
Change in Self-perception of physical fitness | Self-perception of physical fitness will be assessed at week 0 (pre-intervention) and week 13 (post-intervention).
  This assessment will be obtained through the International Fitness Scale - IFIS. The instrument consists of five questions, where higher scores indicate better self-perceptions of physical fitness.
Change in Cognitive failures | Cognitive failures will be assessed at week 0 (pre-intervention) and week 13 (post-intervention).
  This assessment will be obtained through the Questionnaire of Cognitive Flaws (QCF). The instrument consists of 25 questions, and the results are verified through the sum of each of the answered items, ranging from 0 to 100. High scores indicate greater behavioral errors caused by cognitive distortions.
Change in Strength | Strength will be assessed at week 0 (pre-intervention) and week 13 (post-intervention).
  This assessment will be obtained through the hand grip by a hydraulic dynamomete. The higher the values verified in the test, the greater strength.
Change in Power | Power will be assessed at week 0 (pre-intervention) and week 13 (post-intervention).
  This assessment will be obtained through the Power of lower limbs will be evaluated through the horizontal jump test. The higher the values verified in the test, the greater power.
Change in Endurance Strength | Endurance strength will be assessed at week 0 (pre-intervention) and week 13 (post-intervention).
  This assessment will be obtained through the Endurance strength and will be measured by the 1-minute abdominal endurance test. The higher the values verified in the test, the greater endurance strength.
Change in Cardiorespiratory Fitness | Cardiorespiratory Fitness will be assessed at week 0 (pre-intervention) and week 13 (post-intervention).
  This assessment will be obtained through the 20m back and forth test. The higher the values verified in the tests through the distance traveled, in meters, the greater the estimates of maximum oxygen consumption.

REFERENCES:
- [Background] ASHDOWN-FRANKS, G.; SABISTON, C.M.; SOLOMON-KRAKUS, S.; O'LOUGHLIN, J.L. Sport participation in high school and anxiety symptoms in young adulthood. Ment Health Phys Act. 2017;12:19-24.
- [Background] Bordoni B, Purgol S, Bizzarri A, Modica M, Morabito B. The Influence of Breathing on the Central Nervous System. Cureus. 2018 Jun 1;10(6):e2724. doi: 10.7759/cureus.2724. PMID 30083485
- [Background] Broadbent DE, Cooper PF, FitzGerald P, Parkes KR. The Cognitive Failures Questionnaire (CFQ) and its correlates. Br J Clin Psychol. 1982 Feb;21(1):1-16. doi: 10.1111/j.2044-8260.1982.tb01421.x. PMID 7126941
- [Background] Busch V, Magerl W, Kern U, Haas J, Hajak G, Eichhammer P. The effect of deep and slow breathing on pain perception, autonomic activity, and mood processing--an experimental study. Pain Med. 2012 Feb;13(2):215-28. doi: 10.1111/j.1526-4637.2011.01243.x. Epub 2011 Sep 21. PMID 21939499
- [Background] Chen YF, Huang XY, Chien CH, Cheng JF. The Effectiveness of Diaphragmatic Breathing Relaxation Training for Reducing Anxiety. Perspect Psychiatr Care. 2017 Oct;53(4):329-336. doi: 10.1111/ppc.12184. Epub 2016 Aug 23. PMID 27553981
- [Background] Cole TJ, Lobstein T. Extended international (IOTF) body mass index cut-offs for thinness, overweight and obesity. Pediatr Obes. 2012 Aug;7(4):284-94. doi: 10.1111/j.2047-6310.2012.00064.x. Epub 2012 Jun 19. PMID 22715120
- [Background] FERNÁNDEZ-RÍO, J. Another step in models-based practice: Hybridizing Cooperative Learning and Teaching for Personal and Social Responsibility. J Phys Educ Recreat Danc. 2014;85(7):3-5.
- [Background] FERNÁNDEZ-RIO, J.M.; MÉNDEZ-GIMÉNEZ, A. El Aprendizaje Cooperativo: Modelo Pedagógico para Educación Física (Cooperative learning: Pedagogical Model for Physical Education). Retos. 2016;2041(29):201-6.
- [Background] FERNÁNDEZ-RIO, J.; CALDERÓN, A.; HORTIGÜELA ALCALÁ, D.; PÉREZ PUEYO, Á.; AZNAR CEBAMANOS, M. Modelos pedagógicos en Educación Física: consideraciones teórico-prácticas para docentes. Rev Española Educ Física y Deport REEFD. 2016;(413):55-75.
- [Background] Fleck MP, Louzada S, Xavier M, Chachamovich E, Vieira G, Santos L, Pinzon V. [Application of the Portuguese version of the abbreviated instrument of quality life WHOQOL-bref]. Rev Saude Publica. 2000 Apr;34(2):178-83. doi: 10.1590/s0034-89102000000200012. Portuguese. PMID 10881154
- [Background] Foster C. Monitoring training in athletes with reference to overtraining syndrome. Med Sci Sports Exerc. 1998 Jul;30(7):1164-8. doi: 10.1097/00005768-199807000-00023. PMID 9662690
- [Background] GARCÍA, F.; MUSITU, G. Manual Af-5. Autoconcepto forma 5. Madrid: TEA; 2014.
- [Background] Gomez-Baya D, Calmeiro L, Gaspar T, Marques A, Loureiro N, Peralta M, Mendoza R, Gaspar de Matos M. Longitudinal Association between Sport Participation and Depressive Symptoms after a Two-Year Follow-Up in Mid-Adolescence. Int J Environ Res Public Health. 2020 Oct 14;17(20):7469. doi: 10.3390/ijerph17207469. PMID 33066534
- [Background] Heijnen S, Hommel B, Kibele A, Colzato LS. Neuromodulation of Aerobic Exercise-A Review. Front Psychol. 2016 Jan 7;6:1890. doi: 10.3389/fpsyg.2015.01890. eCollection 2015. PMID 26779053
- [Background] Kraemer WJ, Ratamess NA. Fundamentals of resistance training: progression and exercise prescription. Med Sci Sports Exerc. 2004 Apr;36(4):674-88. doi: 10.1249/01.mss.0000121945.36635.61. PMID 15064596
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Kieling C, Baker-Henningham H, Belfer M, Conti G, Ertem I, Omigbodun O, Rohde LA, Srinath S, Ulkuer N, Rahman A. Child and adolescent mental health worldwide: evidence for action. Lancet. 2011 Oct 22;378(9801):1515-25. doi: 10.1016/S0140-6736(11)60827-1. Epub 2011 Oct 16. PMID 22008427
- [Background] Leger LA, Lambert J. A maximal multistage 20-m shuttle run test to predict VO2 max. Eur J Appl Physiol Occup Physiol. 1982;49(1):1-12. doi: 10.1007/BF00428958. PMID 7201922
- [Background] MATSUDO, S.; ARAÚJO, T.; MATSUDO, V.; ANDRADE, D.; ANDRADE, E.; OLIVEIRA, L.; et al. Questionário Internacional de Atividade Física (IPAQ): Estudo De Validade e Reprodutibilidade No Brasil. Rev Bras Atividade Física Saúde. 2001;6(2):5-18.
- [Background] Pascoe MC, Parker AG. Physical activity and exercise as a universal depression prevention in young people: A narrative review. Early Interv Psychiatry. 2019 Aug;13(4):733-739. doi: 10.1111/eip.12737. Epub 2018 Oct 10. PMID 30302925
- [Background] Poirel E. [Psychological benefits of physical activity for optimal mental health]. Sante Ment Que. 2017 Spring;42(1):147-164. French. PMID 28792566
- [Background] Roberts HC, Denison HJ, Martin HJ, Patel HP, Syddall H, Cooper C, Sayer AA. A review of the measurement of grip strength in clinical and epidemiological studies: towards a standardised approach. Age Ageing. 2011 Jul;40(4):423-9. doi: 10.1093/ageing/afr051. Epub 2011 May 30. PMID 21624928
- [Background] SARRIERA, J.C.; CASAS, F.; BEDIN, L.M.; ABS, D.; DOS SANTOS, B.R.; BORGES, F.C.; et al. Propriedades psicométricas da Escala de Autoconceito Multidimensional em adolescentes brasileiros. Aval Psicol. 2015;14(2):281-90.
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Wassenaar TM, Wheatley CM, Beale N, Nichols T, Salvan P, Meaney A, Atherton K, Diaz-Ordaz K, Dawes H, Johansen-Berg H. The effect of a one-year vigorous physical activity intervention on fitness, cognitive performance and mental health in young adolescents: the Fit to Study cluster randomised controlled trial. Int J Behav Nutr Phys Act. 2021 Mar 31;18(1):47. doi: 10.1186/s12966-021-01113-y. PMID 33789683
- [Background] Werner-Seidler A, Perry Y, Calear AL, Newby JM, Christensen H. School-based depression and anxiety prevention programs for young people: A systematic review and meta-analysis. Clin Psychol Rev. 2017 Feb;51:30-47. doi: 10.1016/j.cpr.2016.10.005. Epub 2016 Oct 24. PMID 27821267
- [Background] WORLD HEALTH ORGANIZATION. Depression and other common mental disorders. Global health estimates. WHO; 2017.